CLINICAL TRIAL: NCT05771545
Title: Telepsychiatry to Enable Expedited Disposition of Psychiatric Emergencies
Status: Active, not recruiting | Type: Observational
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Adam Rose, Associate Professor, Hebrew University of Jerusalem
Other Study IDs: HebrewUJ123
Record Dates: First submitted 2023-03-02; First posted 2023-03-16 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Psychiatric Emergency
Keywords: telepsychiatry; implementation science

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Innovation (Usual Care): Patients evaluated in the psychiatric emergency department for possible involuntary admission during the year prior to the innovation in care. During this period, the attending psychiatrist was required to physically come to the hospital to examine the patient.
- Innovation (Tele-Psychiatry): Patients evaluated in the psychiatric emergency department for possible involuntary admission during the innovation period. Instead of physically coming to the hospital, the attending physician will evaluate the patient via video-link, which will be facilitated by the on-site psychiatric resident.
  Interventions: Other: Telepsychiatry

INTERVENTIONS:
Other: Telepsychiatry — Instead of coming to the hospital physically, the attending psychiatrist will evaluate the patient via a video-link.
  Groups: Innovation (Tele-Psychiatry)

SUMMARY:
The goal of this observational study is to examine the effect of using a video link for evaluation of patients in the psychiatric emergency room. Under current Israeli law, the attending physician must come in to physically examine the patient before they can be admitted involuntarily. Patients often de-compensate and even may become violent while waiting for the attending to arrive. Previous studies have shown that evaluation of such patients via video-link has an extremely high concordance with in person evaluation. This study will compare patients who are evaluated via video-link with historical controls evaluated under usual conditions. This is an observational study, which is taking advantage of a change in practice to collect data on two different ways of delivering care, via chart reviews. If successful, this study will show that the video-link is feasible and acceptable to patients and staff. The following hypotheses will be tested:

1. The intervention will result in shorter ED time compared to historical controls.
2. The intervention will result in fewer violent incidents compared to historical controls.
3. The intervention will result in shorter overall hospital length of stay compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Must be evaluated in the psychiatric ED for potential involuntary admission

Exclusion Criteria:

* Not justice-involved (i.e., brought in by police after committing a crime)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are evaluated for involuntary psychiatric admission via the ED, who meet the above criteria.
Sampling Method: Non-Probability Sample
Enrollment: 959 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (8):
- Israel (8):
  - HaEmek Medical Center, Afula
  - Jerusalem Mental Health Center - Eitanim, Jerusalem
  - Jerusalem Mental Health Center, Jerusalem
  - Shaar Menashe Psychiatric Hospital, Pardés H̱anna Karkur
  - Geha Psychiatric Hospital, Petah Tikva
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Lev Hasharon Mental Health Center, Tsur Moshe

IPD SHARING:
Plan to Share IPD: No
It is not possible to share IPD because of data security concerns and the stipulations of the research ethics committees that are approving the study

REFERENCES:
- [Derived] Shalev L, Bistre M, Lubin G, Avirame K, Raskin S, Linkovski O, Eitan R, Rose AJ. Enabling Expedited Disposition of Emergencies Using Telepsychiatry in Israel: Protocol for a Hybrid Implementation Study. JMIR Res Protoc. 2023 Oct 17;12:e49405. doi: 10.2196/49405. PMID 37847548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-Innovation (Usual Care) | Innovation (Tele-Psychiatry)
Started | 525 | 434
Completed | 525 | 434
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Innovation (Usual Care) | Innovation (Tele-Psychiatry) | Total
Number analyzed (Participants) | 525 | 434 | 959
Age, Customized [Count of Participants; unit: Participants]
  Age 18-33 | 226 | 205 | 431
  Age 34-50 | 175 | 129 | 304
  Age 51-68 | 88 | 76 | 164
  Age 69+ | 36 | 24 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 161 | 364
  Male | 322 | 273 | 595
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Jewish | 443 | 377 | 820
  Arab | 76 | 56 | 132
  Foreign Workers or Tourists | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  Israel | 525 | 434 | 959

OUTCOME MEASURES:

1. Primary Outcome: ED Time
Description: Amount of time, in hours and minutes, that the patient spends in the ED prior to disposition
Time Frame: Patients arrive in the ED at a specific time and leave the ED at a specific time. We will compute the amount of time spent in the ED by each patient, up to two weeks.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Pre-Innovation (Usual Care) | Innovation (Tele-Psychiatry)
Number analyzed (Participants) | 525 | 434
Minutes | 106 [70 to 159] | 103 [65 to 155]

2. Secondary Outcome: Violent Incidents
Description: Adjudicated violent incidents that occur, whether in the ED or on the psychiatry ward. Includes hitting, kicking, throwing, and property destruction
Time Frame: Patients arrive in the ED at a specific time. Those who are admitted are eventually discharged. Violent incidents can occur during the entire time spent in the hospital, whether in the ED or on the ward, up to 90 days total.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Innovation (Usual Care) | Innovation (Tele-Psychiatry)
Number analyzed (Participants) | 525 | 434
Participants | 108 | 96

3. Secondary Outcome: Hospital Length of Stay
Description: Length of stay, in days, starting with time of arrival to ED
Time Frame: For patients admitted to the hospital through the ED, the beginning time is their arrival to ED, the end is the time of hospital discharge, up to 90 days later.
Population: Only those who were admitted to hospital; does not include those discharged from the Emergency Department
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pre-Innovation (Usual Care) | Innovation (Tele-Psychiatry)
Number analyzed (Participants) | 388 | 343
days | 18 [9 to 39] | 23 [11 to 41]

ADVERSE EVENTS:
Time Frame: Through hospital discharge or discharge from the emergency department
Arm/Group | Pre-Innovation (Usual Care) | Innovation (Tele-Psychiatry)
All-Cause Mortality (participants affected / at risk) | 0/525 | 0/434
Serious Adverse Events (participants affected / at risk) | 0/525 | 0/434
Other Adverse Events (participants affected / at risk) | 0/525 | 0/434

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT05771545/Prot_SAP_000.pdf